CLINICAL TRIAL: NCT07406516
Title: Identification of Kinematic Variables Specific of Patellar Tendinopathy in Athletes at Risk
Acronym: TENVOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL25_0117; 2025-A01948-41 (Registry Identifier: IdRCB)
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Patellar Tendinitis; Jumper's Knee; Musculoskeletal Injuries; Knee Injuries
Keywords: patellar tendinopathy; injury; Jumper's knee; Biomechanical variables; Biomechanical modeling; Measurement in an ecological environment; Profiling; Markerless technology
MeSH Terms: conditions — Knee Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patellar tendinopathy group (Experimental): Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology.
  Interventions: Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology.
- healthy group (Other): Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology.
  Interventions: Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology at 6 months and 12 months

INTERVENTIONS:
Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology. — Participants will undergo clinical evaluations including the Single Leg Decline Squat (SLDS) test, VISA-PF, OSTRC-P questionnaires, and Doppler ultrasound of the patellar tendon. These assessments will take place at baseline (T0) and follow-up periods (M3, M6, M9, M12) to track the evolution of kinematic markers and clinical symptoms related to patellar tendinopathy.
  Arms: patellar tendinopathy group
Diagnostic Test: The intervention consists of a series of vertical jump tests captured using high-resolution cameras with markerless motion capture technology at 6 months and 12 months — Participants will undergo clinical evaluations including the Single Leg Decline Squat (SLDS) test, VISA-PF, OSTRC-P questionnaires, and Doppler ultrasound of the patellar tendon. These assessments will take place at baseline (T0) and follow-up periods ( M6 et M12) to track the evolution of kinematic markers and clinical symptoms related to patellar tendinopathy.
  Arms: healthy group

SUMMARY:
This research aims to identify and monitor specific kinematic markers associated with patellar tendinopathy in athletes at risk. Using a markerless motion capture system, vertical jump tests will be analyzed to detect early biomechanical changes in the knees, hips, trunk, and ankles. By comparing injured participants, the study seeks to improve early diagnosis and personalized prevention strategies for patellar tendinopathy.

DETAILED DESCRIPTION:
Patellar tendinopathy, also known as Jumper's knee, is the most common pathology in elite sports, with 30% of diagnoses occurring in volleyball. Among elite volleyball players, the prevalence of this overuse-related condition ranges between 40% and 50%, resulting in anterior knee pain during daily and recreational activities, which can lead to deficits in strength and sports performance. To date, investigator can determine whether a patient has had a history of tendinopathy through modifications in biomechanical jump-landing strategies. However, there is a lack of early biomechanical markers to identify the onset of patellar tendinopathy and thus prevent its chronic progression. A preventive strategy using markerless motion capture technology, providing quantitative and visual feedback of a 3D human body model, shows promise. Investigators hypothesize that jump-landing kinematic analysis using markerless technology could identify early kinematic markers specific to patellar tendinopathy, distinguishing affected individuals from a non-tendinopathy population. This could ultimately help identify motor strategies following the onset of patellar tendinopathy A prospective longitudinal multicenter cohort. After signing the consent form, participants will undergo a medical examination, including a clinical assessment, a SLDS test, a Doppler ultrasound of the patellar tendon, and evaluation using the VISA-PF and OSTRC-P scores. Following a standardized 10-minute warm-up, participants will perform vertical jump tests captured by high-resolution cameras, analyzed using markerless motion capture technology. These assessments will be conducted at inclusion and at 3, 6, 9, and 12 months. Additional medical visits will occur if symptoms arise outside of testing.

ELIGIBILITY:
* Subject aged between 18 and 45 years
* Male subject
* Regularly participating in physical activity involving jumping (a predisposing factor for patellar tendinopathy) twice a week for at least one year.
* Participants affiliated with or covered by a social security scheme

SPECIFIC INCLUSION CRITERIA FOR THE PATELLAR TENDINOPATHY GROUP

Patients with at least 2 of the following 3 criteria:

* Modified Öhberg score ≥2 according to L Öhberg, H Alfredson (2002)
* VISA-PF < 80/100 according to Kaux et al. (2016) and/or OSTRC P ≥ 6/100 according to Owoeye et al. (2018)
* Single Leg Decline Squat (SLDS): VAS ≥ 1/10 with pain mapping at the patellar tendon; according to Coombes et al. (2020)

SPECIFIC INCLUSION CRITERIA FOR THE HEALTHY GROUP

Patients with 0 or 1 of the following 3 criteria:

* Modified Öhberg score ≥2 according to L Öhberg, H Alfredson (2002)
* VISA-PF < 80/100 according to Kaux et al. (2016) and/or OSTRC P ≥ 6/100 according to Owoeye et al. (2018)
* Single Leg Decline Squat (SLDS): VAS ≥ 1/10 with pain mapping at the patellar tendon; according to Coombes et al. (2020)

Non inclusion Criteria:

* Significant medical and surgical history involving the lower limbs (e.g., ACL ligament reconstruction, meniscectomy, etc.)
* Contraindications to participating in sports activities
* Other pathologies involving the lower limbs (< 6 months), e.g., torn knee ligaments, ankle sprain, knee sprain, etc.
* Participants who have not given their informed consent
* Participants subject to legal protection measures (legal guardianship, conservatorship, curatorship)
* Participants deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Variations of knee flexion angle at initial contact at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of knee flexion angle at initial contact at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of knee flexion angle at initial contact at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of knee flexion angle at initial contact at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum knee flexion angle at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum knee flexion angle at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum knee flexion angle at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum knee flexion angle at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the knee between initial contact and maximum flexion angle at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the knee between initial contact and maximum flexion angle at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the knee between initial contact and maximum flexion angle at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the knee between initial contact and maximum flexion angle at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF)at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Comparison of variation between healthy group and patellar tendinopathy group of knee flexion angle at initial contact at 6 months | Between the two 6-month visits of the two groups
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Comparison between the healthy group and the patellar tendinopathy group of variation of the maximum knee flexion angle at 6 months | Between the two 6-month visits of the two groups
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Comparison between the healthy group and the patellar tendinopathy group of variations of the range of motion (ROM) of the knee between initial contact and maximum flexion angle at 6 months | Between the two 6-month visits of the two groups
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Comparison between the healthy group and the patellar tendinopathy group of variations of the angle at the peak of the vertical ground reaction force (VGRF)at 6 months | Between the two 6-month visits of the two groups
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.

SECONDARY OUTCOMES:
Variations of the angle of flexion of the trunk, hips, knees, and ankles at initial contact at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle of flexion of the trunk, hips, knees, and ankles at initial contact at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle of flexion of the trunk, hips, knees, and ankles at initial contact at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle of flexion of the trunk, hips, knees, and ankles at initial contact at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum flexion angle of the trunk, hips, knees, and ankles upon landing at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum flexion angle of the trunk, hips, knees, and ankles upon landing at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum flexion angle of the trunk, hips, knees, and ankles upon landing at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the maximum flexion angle of the trunk, hips, knees, and ankles upon landing at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the trunk, hips, knees, and ankles between initial contact and maximum flexion angle upon landing at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the trunk, hips, knees, and ankles between initial contact and maximum flexion angle upon landing at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the trunk, hips, knees, and ankles between initial contact and maximum flexion angle upon landing at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the range of motion (ROM) of the trunk, hips, knees, and ankles between initial contact and maximum flexion angle upon landing at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) of the hips, knees, and ankles upon landing at 3 months (only for patients in the patellar tendinopathy group) | Between the initial visit and the 3-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) of the hips, knees, and ankles upon landing at 6 months | Between the 3-month visit and the 6-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) of the hips, knees, and ankles upon landing at 9 months (only for patients in the patellar tendinopathy group) | Between the 6-month visit and the 9-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.
Variations of the angle at the peak of the vertical ground reaction force (VGRF) of the hips, knees, and ankles upon landing at 12 months | Between the 9-month visit and the 12-month visit
  The participant will perform the required vertical jump tests. The kinematic data will be captured by the investigating physical therapist specializing in motion analysis using a camera and markerless technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Sports Medicine and Traumatology LAPEYRONIE Hospital - Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided